CLINICAL TRIAL: NCT06627660
Title: Manual Valsalva Maneuver As a Preventive Measure of Postoperative Laryngospasm in Laryngomalacia Cases Undergoing Supraglottoplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sameh Fathy (Other)
Responsible Party: Sponsor-Investigator, Sameh Fathy, Sameh Mohamed Fathy El-Sherbiny, MD, Assistant Professor at Mansoura Faculty of Medicine, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Valsalva for laryngospasm
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Laryngomalacia; Laryngospasm
Keywords: VALSALVA MANEUVER; Postoperative Laryngospasm; Supraglottoplasty
MeSH Terms: conditions — Laryngomalacia; Laryngismus | interventions — Valsalva Maneuver

STUDY DESIGN:
Intervention Model Description: INTERVENTIONAL
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group C (No Intervention): Control group
- Group V (Active Comparator): Repeated Valsalva maneuver will be done after recovery from anesthesia
  Interventions: Procedure: Valsalva maneuver

INTERVENTIONS:
Procedure: Valsalva maneuver — Closure of the nose and mouth during expiration for 20 sec
  Arms: Group V

SUMMARY:
We hypothesized that manual valsalva maneuver prevent incidence of postoperative laryngospasm after supraglottoplasty for cases of congenital laryngomalacia.

Primary outcome: Incidence of postoperative stridor and laryngospasm Secondary outcome: incidence of reintubation, postoperative hemodynamics, duration of postoperative ICU and hospital stay

DETAILED DESCRIPTION:
Congenital Laryngomalacia is the main cause of stridor in newborns and infants, affecting 45-75% of all infants with congenital stridor. Short aryepiglottic folds, redundant arytenoid, omega-shaped epiglottis, and inspiratory stridor are features of laryngomalacia. Pediatric laryngospasm is a glottic closure due to reflex constriction of the laryngeal muscles that produce partial or complete obstruction of the larynx. When complete and sustained, laryngospasm is considered an anesthetic Emergency.

The valsalva maneuver involves expiratory effort against a closed glottis in the sitting or supine position with the intraoral and intrathoracic pressures raised to 40 mmHg for 15-20 sec, after which the pressure is suddenly released and the breathing restored to normal.

We hypothesized that manual valsalva maneuver prevent incidence of postoperative laryngospasm after supraglottoplasty for cases of congenital laryngomalacia.

After approval of IRB, Mansoura University, this study will be conducted on infants and children ASA I or II aging from 1 month age- 6 years undergoing supraglottoplasty in Mansoura university hospitals. After obtaining a written informed consent from patients parents, random number generator with closed envelope technique will randomize patients into two groups [control] group ( C group ), Valsalva group ( V group)].

Anesthesia will be induced by inhalational induction using sevoflurane at concentration (6:8%). After that, a proper sized cannula will be introduced with giving atropine 0,01mg/kg and hydrocortisone 4mg/ kg. Then, patients will be seen by fiberoptic endoscopy by the surgeon to detect the stage of laryngomalacia and the supraglottic pathology. After that, proper sized ETT will be inserted using succinylcholine 1mg\kg IV and fixed in place after confirmation of correct positioning , with maintenance of anesthesia with isoflurane. All patients will be given 0.5-1mic /kg fentanyl and 15 mg /kg paracetamol.

A pilot study will be done including 5 patients in each study group. The Incidence of postoperative stridor will be used as the primary variable with difference between studied groups was 40% (50% in group C versus 10% in group V). G*power software version 3.1.9.2 will be utilized to detect the required sample size for a study power of 90% and alpha error of 0.05. Cases involved in the pilot study will not be included in the total sample size of the study. Then total sample size will be 26 in each group and by adding 10% to compensate for possible drop out then total sample size per group will be 29 cases in each group. Perioperative data will be tabulated and analyzed using IBM SPSS software version 26.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children ASA I or II aging from 1 month age - 6 years undergoing supraglottoplasty

Exclusion Criteria:

* Parents refusal.
* Patients with increased ICP
* Patients with increased IOP

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2024-10-06 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of laryngospasm | 24 HOURS

SECONDARY OUTCOMES:
incidence of reintubation | 24 HOURS
Postoperative oxygen saturation measurement | 1 HOUR
  Oxygen saturation (%) is recorded every 5 minutes
Incidence of postoperative nausea and vomiting | 24 HOURS
Duration of postoperative hospital stay | 24 HOURS

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshahat Aboelfoutouh, DOCTORAL DEGREE (MD), Principal Investigator — Lecturer of Anesthesia and Surgical Intensive Care - Faculty of medicine - Mansoura university; Rania Elmohamady Elbadrawy, DOCTORAL DEGREE (MD), Principal Investigator — Lecturer of Anesthesia and Surgical Intensive Care- Faculty of medicine - Mansoura university

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kumar CM, Van Zundert AAJ. Intraoperative Valsalva maneuver: a narrative review. Can J Anaesth. 2018 May;65(5):578-585. doi: 10.1007/s12630-018-1074-6. Epub 2018 Jan 24. PMID 29368315
- [Background] Ramprasad VH, Ryan MA, Farjat AE, Eapen RJ, Raynor EM. Practice patterns in supraglottoplasty and perioperative care. Int J Pediatr Otorhinolaryngol. 2016 Jul;86:118-23. doi: 10.1016/j.ijporl.2016.04.039. Epub 2016 May 3. PMID 27260594
- [Background] Alalami AA, Ayoub CM, Baraka AS. Laryngospasm: review of different prevention and treatment modalities. Paediatr Anaesth. 2008 Apr;18(4):281-8. doi: 10.1111/j.1460-9592.2008.02448.x. PMID 18315632
- [Background] Hernández-Cortez E. Update on the management of laryngospasm. J Anesth Crit Care Open Access. 2018;8(2):1-6.
- [Background] Birlie Chekol W, Yaregal Melesse D. Incidence and Associated Factors of Laryngospasm among Pediatric Patients Who Underwent Surgery under General Anesthesia, in University of Gondar Compressive Specialized Hospital, Northwest Ethiopia, 2019: A Cross-Sectional Study. Anesthesiol Res Pract. 2020 Jan 24;2020:3706106. doi: 10.1155/2020/3706106. eCollection 2020. PMID 32411216
- [Background] Oshan V and Robert WM. Anesthesia for complex airway surgery in children. Continuing Education in Anesthesia, Critical care and Pain 2013;13:47-51